CLINICAL TRIAL: NCT03161821
Title: Quantification and Characterization of Circulating Tumor Cells in Solid Tumors
Brief Title: Circulating Tumor Cells in Solid Tumors
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1121; 11-1924 (Other: UNC IRB)
Record Dates: First submitted 2017-05-15; First posted 2017-05-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational

SUMMARY:
The purpose of this study is to identify circulating tumor cells in patients with solid tumors. Quantify and characterize these cells, collect patient information in regards to the patient's cancer. Develop a database and a sample repository where future analysis could be done.

DETAILED DESCRIPTION:
The primary purpose of this correlative study is to create a prospective database documenting the quantity and characterization of circulating tumor cells (CTCs) in solid tumor patients as identified by a various laboratory techniques and analyses. The investigators are developing this resource to provide data to achieve the following objectives: 1) correlate CTCs with known prognostic factors, 2) correlate CTCs with burden of disease, 3) evaluate the ability of CTCs to be used in the surveillance of disease recurrence, and 4) evaluate CTCs ability to be used as a biomarker for treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Biopsy proven solid tumor malignancy
* Seen at UNC Chapel Hill Hospital and Health Care System
* Consents to abstraction of their medical records
* Signed an institutional review board (IRB)-approved informed consent document for this protocol

Exclusion Criteria:

* < 18 years of age
* Dementia, altered mental status, incarceration or any psychiatric condition that would prohibit the understanding or rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancerous solid tumors
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2011-12-09 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Documentation of the Quality of CTCs from Patients with Solid Tumors | Through study completion, an average of 5 years
  Enumeration of participants' circulating solid tumor cells
Documentation of the Characterization of CTCs from Patients with Solid Tumors | Through study completion, an average of 5 years
  Characterization of participants' circulating solid tumor cells

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Carey, MD, Principal Investigator — University of North Carolina
Locations (1):
- Radiation Oncology Clinic - UNC Cancer Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chera BS, Kumar S, Shen C, Amdur R, Dagan R, Green R, Goldman E, Weiss J, Grilley-Olson J, Patel S, Zanation A, Hackman T, Blumberg J, Patel S, Thorp B, Weissler M, Yarbrough W, Sheets N, Mendenhall W, Tan XM, Gupta GP. Plasma Circulating Tumor HPV DNA for the Surveillance of Cancer Recurrence in HPV-Associated Oropharyngeal Cancer. J Clin Oncol. 2020 Apr 1;38(10):1050-1058. doi: 10.1200/JCO.19.02444. Epub 2020 Feb 4. PMID 32017652
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials